CLINICAL TRIAL: NCT01294553
Title: An Open Label, Multi-centre, Non-interventional Post-marketing Surveillance to Monitor the Safety and/or Efficacy of Avandamet® Administered in Korean Diabetic Patients According to the Prescribing Information
Brief Title: An Open Label, Multi-centre, Non-interventional Post-marketing Surveillance to Monitor the Safety and/or Efficacy of AVANDAMET Between June 2004 and January 2010
Acronym: AVANDAMETPMS
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 105709
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Results first posted 2011-03-15 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2011-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- rosiglitazone/metformin group: Korean subjects who are administered rosiglitazone/metformin according to the prescription information
  Interventions: Drug: Administration of rosiglitazone/metformin

INTERVENTIONS:
Drug: Administration of rosiglitazone/metformin — Subjects who are administered rosiglitazone/metformin at least once
  Other Names: according to label and physician's decision based on each subject's condition

SUMMARY:
An open label, multi-centre, non-interventional post-marketing surveillance to monitor the safety and/or efficacy of rosiglitazone/metformin administered in Korean Diabetic patients according to the prescribing information

DETAILED DESCRIPTION:
An open label, multi-centre, non-interventional post-marketing surveillance to monitor the safety and/or efficacy of rosiglitazone/metformin administered in Korean Diabetic patients according to the prescribing information

ELIGIBILITY:
Inclusion criteria

* Subjects administered with rosiglitazone/metformin as an adjunct to diet and exercise for the treatment of type2 diabetes mellitus
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol and follow the administration regimen
* Subjects administered with rosiglitazone/metformin following the locally approved prescribing information

Exclusion criteria

* Subjects with previous history of hypersensitivity to rosiglitazone and/or metformin or any other ingredient
* Subjects with previous history of lactic acidosis, renal disease or renal dysfunction, hepatic dysfunction, cardiogenic shock, heart failure, myocardial infarction, pulmonary infarction and any other status with stomach upset
* Subjects with type 1 diabetes mellitus
* Subjects with acute or chronic metabolic acidosis, including diabetic ketoacidosis, with or without coma
* Subjects with severe infection, pre/post surgery, severe trauma
* Subjects with malnutrition, inanition, emaciation, pituitary insufficiency, adrenal insufficiency
* Subjects undergoing radiologic studies involving intravascular administration of iodinated contrast materials

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type II diabets mellitus patients prescribed rosiglitazone/metformin in general hospital
Sampling Method: Probability Sample
Enrollment: 717 (Actual)
Dates: Start 2004-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The objective of this post-marketing surveillance (PMS) study was to monitor the safety and efficacy of Avandamet in the real clinical setting after launch.
Groups:
- Avandamet 1/500, 2/500, 4/500, 2/1000, or 4/1000 mg: Participants were assigned to the appropriate dose of Avandamet tablet based on their current regimen (fixed dose combination of rosiglitazone and metformin, 1/500 milligrams [mg], 2/500 mg, 4/500 mg, 2/1000 mg, or 4/1000 mg). Participants were not to have exceeded the maximum recommended daily dose of 8/2000. All participants were to have started the rosiglitazone component of Avandamet at the lowest recommended dose, and all dose increases should have been accompanied by careful monitoring for adverse events related to fluid retention.
Period: Overall Study
Arm/Group | Avandamet 1/500, 2/500, 4/500, 2/1000, or 4/1000 mg
Started | 982
Completed | 713
Not Completed | 269
Not completed — Duplicated Participants | 1
Not completed — Protocol Violation | 268

BASELINE CHARACTERISTICS:
Groups:
- Avandamet 1/500, 2/500, 4/500, 2/1000, or 4/1000 mg: Participants were assigned to appropriate dose of Avandamet tablet (fixed dose combination of rosiglitazone and metformin, 1/500 milligrams [mg], 2/500 mg, 4/500 mg, 2/1000 mg, or 4/1000 mg) per physician's decision based on participant's condition
Arm/Group | Avandamet 1/500, 2/500, 4/500, 2/1000, or 4/1000 mg
Number analyzed (Participants) | 713
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline characteristics were collected in members of the Intent-to-Treat (ITT) Population, comprised of all participants who had been administered the investigational drug at least once and had undergone all safety assessments.
  Years | 56.4 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline characteristics were collected in members of the ITT population, comprised of all participants who had been administered the investigational drug at least once and had undergone all safety assessments.
  Participants
    Female | 369
    Male | 344
Race/Ethnicity, Customized [Number; unit: participants] — Baseline characteristics were collected in members of the ITT Population, comprised of all participants who had been administered the investigational drug at least once and had undergone all safety assessments.
  participants
    Korean | 713
    Not Korean | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Adverse Event
Description: An adverse event is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. For a list of all adverse events occurring during the course of the study, please see the table entitled "Other (non-serious) adverse events" in the Adverse Event section of the results record.
Time Frame: 41.4 weeks
Population: Intent-to-Treat (ITT) Population: all participants who had been administered the investigational drug at least once and had undergone all safety assessments
Measure: Number; unit: participants
Arm/Group | Avandamet 1/500, 2/500, 4/500, 2/1000, or 4/1000 mg
Number analyzed (Participants) | 713
participants | 110
Statistical Analysis 1: Comparison: Avandamet 1/500, 2/500, 4/500, 2/1000, or 4/1000 mg; Test type: Superiority or Other; Percentage of participants = 15.4, 95% CI 2-sided [12.8 to 18.1] — The estimated value represents the percentage of participants with an adverse event

2. Secondary Outcome: Number of Participants With a Serious Adverse Event
Description: A serious adverse event is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or results in prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect. For a list of all serious adverse events occurring during the course of the study, please see the table entitled "Serious Adverse Events" in the Adverse Event section of the results record.
Time Frame: 41.4 weeks
Population: ITT Population
Measure: Number; unit: participants
Groups:
- Avandamet 1/500, 2/500, 4/500, 2/1000, or 4/1000 mg: Participants were assigned to appropriate dose of Avandamet tablet (fixed dose combination of rosiglitazone and metformin, 1/500 mg, 2/500 mg, 4/500 mg, 2/1000 mg, or 4/1000 mg) per physician's decision based on participant's condition
Arm/Group | Avandamet 1/500, 2/500, 4/500, 2/1000, or 4/1000 mg
Number analyzed (Participants) | 713
participants | 2

3. Secondary Outcome: Number of Participants With the Indicated Unexpected Adverse Events
Description: Unexpected adverse events are defined as those that were not described in the locally approved label by the Korean Food and Drug Administration (KFDA) at the time of surveillance completion.
Time Frame: 41.4 weeks
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Avandamet 1/500, 2/500, 4/500, 2/1000, or 4/1000 mg
Number analyzed (Participants) | 713
participants
  Gastritis | 42
  Dysaesthesia | 5
  Impotence | 3
  Paralysis | 2
  Insomnia | 2
  Depression | 2
  Dermatitis | 2
  Peptic ulcer | 1
  Gastric ulcer | 1
  Temperature changed sensation | 1
  Dermatitis fungal | 1
  Pneumonia | 1
  Skeletal pain | 1
  Osteoporosis | 1
  Myalgia | 1
  Anxiety | 1
  Cystitis | 1
  Renal calculus | 1
  Albuminuria | 1
  Urinary incontinence | 1
  Liver fatty | 1
  Vaginal haemorrhage | 1
  Menopausal symptoms | 1
  Glaucoma | 1
  Coughing | 1
  Exophthalmus | 1
  Teratoma benign | 1
  Cardiomyopathy | 1
  Arteriosclerosis | 1

ADVERSE EVENTS:
Description: Adverse events were coded by using World Health Organization Adverse Reactions Terminology (WHOART, preferred term level) according to the local regulation.
Arm/Group | Avandamet 1/500, 2/500, 4/500, 2/1000, or 4/1000 mg
Serious Adverse Events (participants affected / at risk) | 2/713
Other Adverse Events (participants affected / at risk) | 77/713
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avandamet 1/500, 2/500, 4/500, 2/1000, or 4/1000 mg (N=713)
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Chest pain (General disorders) | 1
Pneumonia (Immune system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Avandamet 1/500, 2/500, 4/500, 2/1000, or 4/1000 mg (N=713)
Upper respiratory tract infection (Immune system disorders) | 17
Oedema (Metabolism and nutrition disorders) | 16
Gastritis (Gastrointestinal disorders) | 9
Weight increase (General disorders) | 8
Dyspepsia (Gastrointestinal disorders) | 6
Headache (General disorders) | 6
Dysaesthesia (Nervous system disorders) | 5
Chest pain (General disorders) | 4
Constipation (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 3
Impotence (Reproductive system and breast disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.